CLINICAL TRIAL: NCT03305965
Title: The Effectiveness of Patient Navigation in Cancer Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N16NVG
Record Dates: First submitted 2017-09-25; First posted 2017-10-10 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: Patient navigation vs. care as usual
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient navigation (Experimental)
  Interventions: Behavioral: Patient navigation
- Care as usual (No Intervention)

INTERVENTIONS:
Behavioral: Patient navigation — Consultations with a specifically trained oncology nurse (i.e. patient navigator), who assesses patients' needs for supportive cancer care, provides information on supportive cancer care, and guides patients through the supportive cancer care system. Consultations with the patient navigator take place at the start, halfway through, and at the end of treatment.
  Arms: Patient navigation

SUMMARY:
Rationale: Supportive care such as physical therapy, psycho-social education, and dietary advice is likely to have a positive effect on the recovery and quality of life of cancer patients. Currently, not all patients know how to access supportive care, which results in unmet supportive care needs. This study determines whether these unmet needs can be reduced or prevented by a patient navigation intervention that focuses on timely screening and systematic monitoring of patient's supportive care needs.

Objective: The primary objective is to determine the effect of patient navigation on health related quality of life. Secondary objectives are: 1) to determine the effect of patient navigation on satisfaction with, need for, and consumption of (supportive) cancer care; 2) to determine the effect of patient navigation on patients' self-management; 3) to explore how patient navigation affects the cost-effectiveness of cancer care.

Study design: Longitudinal randomised controlled trial with two study arms: a patient navigation intervention and care as usual.

Study population: Newly diagnosed lung, melanoma, urology, or gynecology patients of the Netherlands Cancer Institute.

Intervention : Consultations with a specifically trained oncology nurse (i.e. patient navigator), who assesses patients' needs for supportive cancer care, provides information on supportive cancer care, and guides patients through the supportive cancer care system. Consultations with the patient navigator take place at the start, halfway through, and at the end of treatment.

Main study endpoints: The main endpoint of this study is health related quality of life, which is defined as an individual's perceived emotional, social, physical, and functional wellbeing over time. Health related quality of life is assessed with the EORTC QLQ-C30.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants are expected to strongly benefit from consulting the patient navigator without being subjected to any severe risks. Consultations will be provided by highly qualified professionals, and result in benefits such as decreased severity of cancer-related psychosocial and physical distress. To minimise burden, face-to-face consultations will always be scheduled alongside other appointments of at the NKI-AVL. Furthermore, questionnaire completion takes no more than 30 minutes per data collection round, of which three are scheduled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with lung, melanoma, urology or gynecology related cancer
* Male or female
* Treated at the Dutch Cancer Institute
* Has not started treatment at the Dutch Cancer Institute
* 18 years of age and over
* Curative or palliative treatment
* Able to understands and speak Dutch

Exclusion Criteria:

* Not willing to sign the consent form
* Not willing to meet with the patient navigator
* Not willing to complete questionnaires at any point in time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-10-15 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in health related quality of life | Baseline, month 1, month 3, month 5
  EORTC QLQ-C30

SECONDARY OUTCOMES:
Change in need for supportive cancer care | Baseline, month 1, month 3, month 5
  Distress Thermometer
Satisfaction with (supportive) cancer care | Month 5
  (Adapted version of) Patient Satisfaction with Cancer Care
Change in consumption of supportive cancer care | Baseline, month 1, month 3, month 5
  (Adapted version of) Medical Consumption Questionnaire
Change in self-management | Baseline, month 1, month 3, month 5
  Study specific questions on knowledge and self-efficacy
Change in work productivity | Baseline and month 5
  Study specific questions on work productivity
Change in health status | Baseline and month 5
  EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Eveline Bleiker, PhD, Study Director — The Netherlands Cancer Institute
Locations (1):
- Dutch Cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided